CLINICAL TRIAL: NCT07219966
Title: A Phase 3, Multicenter, Randomized, Double-Blind Study to Investigate the Efficacy and Safety of Brenipatide Compared With Placebo for the Treatment of Adult Participants With Moderate-to-Severe Alcohol Use Disorder (RENEW-ALC-1)
Brief Title: A Study of Brenipatide in Participants With Moderate-to-Severe Alcohol Use Disorder
Acronym: RENEW-ALC-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27346; 2025-522313-38-00 (EU CTIS Number); J2S-MC-GZME (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-13; First posted 2025-10-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3537031 Period 1 (Experimental): Escalating doses administered subcutaneously (SC)
  Interventions: Drug: LY3537031; Drug: Placebo
- LY3537031 Period 2 (Experimental): Administered SC
  Interventions: Drug: LY3537031; Drug: Placebo
- Placebo (Placebo Comparator): Administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3537031 — Administered SC
  Other Names: Brenipatide
  Arms: LY3537031 Period 1; LY3537031 Period 2
Drug: Placebo — Administered SC

SUMMARY:
The purpose of this study is to see if brenipatide when compared to a placebo works and is safe for participants with moderate-to-severe Alcohol Use Disorder (AUD). Participation in this study will last approximately 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a minimum of 20 years of age for the investigative sites in Japan.
* Are seeking treatment and are motivated to stop or cut down on drinking.
* Are reliable and willing to make themselves available for the duration of the study and attend required study visits, and are willing and able to follow study procedures as required, such as

  * self-inject study intervention
  * store and use the provided blinded study intervention, as directed
  * maintain electronic and paper study diaries, as applicable, and
  * complete the required questionnaires.

Exclusion Criteria:

* Have evidence of current or within the past 180 days prior to screening (V1), history of any substance use disorder(s) of any severity with a pattern of persistent illicit or nonprescribed substance use as indicated by clinical interview, except alcohol, nicotine, or caffeine.
* Have answered "yes" to either Question 4 or Question 5 on the "Suicidal Ideation" portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) and the ideation occurred within the past 6 months, or have answered "yes" to any of the suicide-related behaviors on the "Suicidal Behavior" portion of the C-SSRS and the behavior occurred within the past 6 months
* Have a history of advanced liver disease (including advanced liver fibrosis or cirrhosis), or alcohol-associated hepatitis based on either prior liver histology or imaging studies, such as transient elastography, ultrasound, computed tomography (CT) and magnetic resonance imaging (MRI), or Enhanced Liver Fibrosis score.
* Have participated in a clinical study and have received active treatment, or unknown if they received active treatment, within 90 days or 5 half-lives (whichever is longer) before screening (V1).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in Drinking Patterns in Alcohol Use Disorder (AUD) as Assessed by the Timeline Followback Method (TLFB) | Up to 56 weeks

SECONDARY OUTCOMES:
Change in Daily Alcohol Consumption as Assessed by the TLFB | Up to 56 weeks
Mean Change in Alcohol Craving as Assessed by the Penn Alcohol Craving Scale (PACS) | Baseline up to Week 56
Mean Change in Alcohol Use Disorders Identification Test (AUDIT) Score | Baseline up to Week 56
Mean Change in Body Weight | Baseline up to Week 56
Mean Change in Patient Reported Health Outcomes as Measured by Short Form 36, v2 (SF-36) Acute Form Domain and Component Summary Scores | Baseline up to Week 56
Pharmacokinetic (PK): Average Steady State Plasma Concentration (Cavg) of Brenipatide | Baseline up to Week 56
Number of Participants with Treatment Emergent Anti-Drug Antibodies (TE-ADA) | Baseline up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (115):
- United States (26):
  - Parkway Medical Center, Birmingham, Alabama
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - UCLA Clinical & Translational Research Center (CTRC), Los Angeles, California
  - Artemis Institute for Clinical Research, San Diego, California
  - UCSF Weill Institute for Neurosciences - Substance Use Disorders Clinic - Mission Bay, San Francisco, California
  - Mountain Mind - Denver, Denver, Colorado
  - Accel Research Sites - Lakeland Clinical Research Unit, Lakeland, Florida
  - K2 Medical Research - Maitland, Maitland, Florida
  - K2 Medical Research ORLANDO, Maitland, Florida
  - Life Arc Research Centers - Miami, Miami, Florida
  - Wellness Research Center, Miami, Florida
  - Life Medical Research Group Corp, Miami Gardens, Florida
  - Charter Research - Orlando, Orlando, Florida
  - K2 Medical Research - Tampa, Tampa, Florida
  - Re:Cognition Health - Chicago, Chicago, Illinois
  - Maryland Treatment Centers - Mountain Manor Treatment Center, Baltimore, Maryland
  - Adams Clinical Bronx, The Bronx, New York
  - North Star Medical Research, Middleburg Heights, Ohio
  - Penn Medicine: University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Avera Research Institute - Sioux Falls, Sioux Falls, South Dakota
  - UT Southwestern Medical Center, Dallas, Texas
  - Adams Clinical Dallas, DeSoto, Texas
  - Pillar Clinical Research - Richardson, Richardson, Texas
  - Alpine Research Organization, Clinton, Utah
  - Re:Cognition Health, Fairfax, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington
- Belgium (5):
  - ANIMA Research, Diepenbeek
  - Kormont, Kluisbergen
  - Gezondheidshuis De Gloed, Machelen
  - Meclinas, Mechelen
  - Medisch Centrum Saffrou, Oudenaarde
- China (27):
  - Beijing Anding Hospital - Affiliated Capital University of Medical Science, Beijing
  - Beijing HuiLongGuan Hospital, Beijing
  - The Second People's Hospital of Hunan Province, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Cheng Du Shi
  - The Fourth People's Hospital of Chengdu, Chengdu
  - Guangzhou Brain Hospital, Guangzhou
  - The Seventh People's Hospital of Hangzhou, Hangzhou
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - The Fourth Hospital of Harbin Medical University, Harbin
  - Huzhou Third Municipal Hospital, Huzhou
  - Shandong Mental Health Center, Jinan
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - The Third Hospital of Mianyang, Mianyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Affilicated Kangning Hospital of Ningbo University, Ningbo
  - Shanghai Mental Health Center, Shanghai
  - Shenzhen Kangning Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - The Affiliated hospital of Southwest Medical University, Sichuan
  - Tianjin Anding Hospital, Tianjin
  - Wuhu Hospital of Beijing Anding hospital, Wuhu
  - Xi An Mental Health Center, Xi'an
  - Xiamen Xianyue Hospital, Xiamen
  - Xianyang Hospital of Yan'an University, Xianyang
  - Psychiatric Hospital of Henan Province, Xinxiang
  - Zhenjiang Mental Health Center, Zhenjiang
- Germany (7):
  - FutureMeds GmbH, Berlin
  - Velocity Clinical Research, Berlin, Berlin
  - Klinische Forschung Dresden, Dresden
  - Klinische Forschung Hamburg, Hamburg
  - Zentralinstitut für Seelische Gesundheit, Mannheim
  - Dedicated Research Site FutureMeds, Offenbach
  - Klinische forschung Schwerin GmbH, Schwerin
- Japan (23):
  - Takahashi Psychiatric Clinic, Ashiya
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Ai Sakura Clinic, Fukuoka
  - Hiro Mental Clinic, Fukuoka
  - Kuramitsu Hospital, Fukuoka
  - Rainbow and Sea Hospital, Karatsu
  - Kariya Hospital, Kariya
  - Tatsuta Clinic, Kobe
  - Arata Clinic, Nagasaki
  - Yokogawa Ekimae Clinic, Nishi
  - Teine Keijinkai Hospital, Sapporo
  - Sangenjaya Shinkeika Shinryonaika Clinic, Setagaya City
  - Hillside Clinic Jingumae, Shibuya City
  - Kaedenomori Mental Clinic, Shibuya City
  - Samoncho Clinic, Shinjuku
  - Keiai Clinic, Shinjuku-ku
  - Higashi Shinjuku Clinic, Shinjuku-ku
  - Sakurazaka Clinic SophyAnce, Tokyo
  - Noguchi Naika Clinic, Tokyo
  - Tsukuba University Hospital, Tsukuba
  - Maekawa Medical Clinic, Yokohama
  - Makoto Kokoro No Clinic, Yokohama
  - National Hospital Organization Hizen Psychiatric Medical Center, Yoshinogari-cho, Kanzaki-gun
- South Korea (13):
  - Pusan National University Yangsan Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Hanyang University Guri Hospital, Guri-si
  - Inha University Hospital, Incheon
  - Kyungpook National University Hospital, Junggu
  - Gachon University Gil Medical Center, Namdong-gu
  - Konyang University Hospital, Seogu
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si
- Taiwan (6):
  - Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City
  - China Medical University Hospital, Taichung
  - Mackay Memorial Hospital, Taipei
  - Taipei City Hospital - Songde Branch, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (8):
  - Charlton Lane, Cheltenham
  - Edinburgh Royal Infirmary, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - St Pancras Clinical Research, London
  - National Institute for Health Research (NIHR) - King's Clinical Research Facility (CRF), London
  - Clerkenwell Health - London - Baker Street, London
  - Salford Royal Hospital, Salford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Brenipatide in Participants With Moderate-to-Severe Alcohol Use Disorder (RENEW-ALC-1) — https://trials.lilly.com/en-US/trial/662497